CLINICAL TRIAL: NCT00547794
Title: AVERT-AF: Atrio-VEntricular Junction Ablation Followed by Resynchronization Therapy in Patients With Congestive Heart Failure and Atrial Fibrillation
Brief Title: AVJ Ablation Followed by Resynchronization Therapy in Patients With CHF and AF
Acronym: AVERT-AF
Status: Terminated | Type: Observational
Why Stopped: Difficulty in patient enrollment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD 310
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation; Congestive Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CRT-D + AVJ Ablation
- Single-Chamber ICD + Pharmacological Therapy

SUMMARY:
The purpose of the study is to determine if the combination of AVJ ablation followed by BiV pacing significantly improves functional status and exercise capacity compared to pharmacologic rate control in patients with chronic AF and depressed ejection fraction, regardless of rate or QRS duration.

DETAILED DESCRIPTION:
* This is a prospective, randomized, double blinded, multicenter study
* Patients meeting all the enrollment criteria are screened at enrollment and randomized to Group 1 (Pharmacological therapy + Single Chamber ICD) or Group 2 (AVJ Ablation + CRT-D)
* Screened patients are implanted with a FDA approved SJM ICD/CRT-D with compatible lead system
* Patients are followed at 1, 3, 6 and 12 months post implant
* Total # of centers - 20 centers
* Sample size - 180 patients

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic permanent AF
* Class I or II indication for ICD
* LVEF ≤ 35% within 6 months
* NYHA class II or III with a history of CHF
* Maximal tolerated drug therapy for CHF and rate control with a stable regimen for ≥ 30 days
* Ability to independently comprehend and complete a QoL questionnaire
* Ability to give informed consent for study participation and willingness and ability to comply with prescribed follow-up tests and scheduled evaluations

Exclusion Criteria:

* Paroxysmal or persistent AF
* Class I indication for pacing (including AVJ ablation for poor rate control)
* Ability to walk ≥ 450 meters in 6 minutes
* Musculoskeletal disorders that prohibit the completion of a 450 meters walk
* NYHA class I or IV at the time of enrollment
* A contraindication to taking Coumadin therapy
* History of myocardial infarction, percutanous coronary intervention, or CABG in the past 30 days
* History of mitral valve surgery
* Prior attempts for cardiac resynchronization therapy
* The presence of an existing coronary sinus lead or epicardial lead
* Life expectancy < 1year
* Age < 18 yrs
* Current participation in other clinical studies except registry trials
* Use of calcium channel blockers
* Pregnancy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with history of permanent AF and CHF
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-06; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Exercise duration | 12 month post implant

SECONDARY OUTCOMES:
Quality of Life (QOL) via Minnesota Living With Heart Failure (MLWH) questionnaire | 12 month post implant
NYHA Class Progression | 12 month post implant
LVEF | 12 month post implant

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamdan, MD, Principal Investigator — University of Utah Health Sciences
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Hamdan MH, Freedman RA, Gilbert EM, Dimarco JP, Ellenbogen KA, Page RL. Atrioventricular junction ablation followed by resynchronization therapy in patients with congestive heart failure and atrial fibrillation (AVERT-AF) study design. Pacing Clin Electrophysiol. 2006 Oct;29(10):1081-8. doi: 10.1111/j.1540-8159.2006.00502.x. PMID 17038140